CLINICAL TRIAL: NCT04521803
Title: IMPI-3 - A Randomized Controlled Trial of High vs. Standard Dose Rifampicin for Effusive Tuberculous Pericarditis
Brief Title: High vs. Standard Dose Rifampicin for Effusive Tuberculous Pericarditis
Acronym: IMPI-3
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cape Town (Other)
Responsible Party: Principal Investigator, Mpiko Ntsekhe, National Principal Investigator, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: IMPI-3 DMID 20-0007
Record Dates: First submitted 2020-07-16; First posted 2020-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-03

CONDITIONS: Tuberculous Pericarditis; HIV Status
MeSH Terms: conditions — Pericarditis, Tuberculous | interventions — Rifampin

STUDY DESIGN:
Intervention Model Description: Participant identification numbers (PID), assigned at the screening visit, will be used throughout the study. After signing the informed consent document; eligible participants will be stratified by HIV status and then further stratified by GX-Ultra status to ensure equal allocation regardless of HIV status and likely subsequent culture status.
  An electronic randomization tool will be used to randomize the subgroups in a 1:1 ratio. The randomization list will be generated and updated by the study coordinator, trial pharmacist, or statistician who will have no direct contact with trial participants or involvement with the assessment for eligibility in the trial.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Neither participants nor the investigators will be aware of the participant's treatment allocation until the end of the study (double blinding). Blinding will be maintained by manufacture of placebo tablets similar in appearance and packaging to that of the study drug, with centralized dispensing by the study pharmacist. Unmasking procedures are detailed by SOP.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Standard of care (RIF10) (No Intervention): Dosing of the daily oral RHZE fixed dose combination (FDC) will be according to WHO weight bands
- Arm 2: High-dose RIF (RIF35) (Experimental): Simulations were performed to determine the dose of RIF required to achieve the most equitable drug exposures across the weight range, 30 to 100 kg. Demographic data of a reference cohort of TB patients (n = 1225), with or without HIV-1 coinfection, recruited in clinical trials conducted in West Africa and South Africa were used for the simulations35-38. An additional 12 250 virtual patients were generated using the weight and height distributions of the 1225 patients to increase the number of patients with a weight close to the boundaries of the weight range. Parameter estimates of the population PK model for RIF were used to simulate (100 replicates) RIF exposures22. Four dosing scenarios were evaluated using the weight-band based dosing with 4-drug FDC tablets and extra RIF tablets with each tablet containing 150 mg or 600 mg RIF. The FDC tablets were assumed to have 20% reduced bioavailability based on data from a clinical trial where the same formulation was used39
  Interventions: Drug: high dose Rifampicin (RIF)

INTERVENTIONS:
Drug: high dose Rifampicin (RIF) — Simulations were performed to determine the dose of RIF required to achieve the most equitable drug exposures across the weight range, 30 to 100 kg. Demographic data of a reference cohort of TB patients (n = 1225), with or without HIV-1 coinfection, recruited in clinical trials conducted in West Africa and South Africa were used for the simulations35-38. An additional 12 250 virtual patients were generated using the weight and height distributions of the 1225 patients to increase the number of patients with a weight close to the boundaries of the weight range. Parameter estimates of the population PK model for RIF were used to simulate (100 replicates) RIF exposures22. Four dosing scenarios were evaluated using the weight-band based dosing with 4-drug FDC tablets and extra RIF tablets with each tablet containing 150 mg or 600 mg RIF. The FDC tablets were assumed to have 20% reduced bioavailability based on data from a clinical trial where the same formulation was used
  Arms: Arm 2: High-dose RIF (RIF35)

SUMMARY:
The investigators hypothesise that high dose RIF (RIF35) will increase pericardial fluid RIF exposure and so enhance mycobacterial clearance, compared to standard of care dosing (RIF10).

This Phase 2b randomized, placebo-controlled, double-blinded trial will evaluate the efficacy and safety of RIF 35mg/kg compared 10mg/kg, added to standard first-line ATT, for the treatment of PCTB.

DETAILED DESCRIPTION:
IMPI-3 - A Randomized Controlled Trial of High vs. Standard Dose Rifampicin for Effusive Tuberculous Pericarditis

Phase 2b Randomized, placebo-controlled, double-blinded clinical trial

The trial will enroll 100 adult participants with pericardial TB from two research sites in South Africa, with no exclusions being made on the basis of sex/gender, racial or ethnic group.

Consenting participants will be stratified by HIV status and PCF GX-Ultra status, then randomized 1:1 to receive either standard of care anti-tuberculosis treatment (ATT) or standard of care plus high dose Rifampicin (RIF), both administered orally for 2 months, followed by a continuation phase of 4 months' RH at standard doses.

ELIGIBILITY:
Inclusion Criteria:

1. Aged >18 years
2. Suspected PCTB with confirmed pericardial effusion on echocardiography (i.e., echo free space of ≥1 cm anterior to the right ventricle in diastole)
3. Consent to study participation including testing for HIV-1 (if HIV status is unknown)
4. Microbiologically detected Mtb in PCF or diagnosis of probable PCTB. Probable PCTB (in the absence of a positive pericardial fluid culture) will be defined as per Mayosi et al.4:

   1. Evidence of pericarditis with microbiologic confirmation of Mtb- infection elsewhere in the body and/or
   2. Exudative, lymphocyte predominant effusion with elevated adenosine deaminase (≥35 U/L)
5. Participant will undergo pericardiocentesis (as per clinical indication)
6. Within 5 days of ATT initiation

Exclusion Criteria:

1. Glomerular filtration rate <30ml/min or renal failure requiring dialysis
2. Rifampin-resistant TB
3. Severe concurrent opportunistic infection
4. Contraindication to placement of intra-pericardial catheter
5. Failed pericardiocentesis procedure and/or failure of placement of intra-pericardial catheter
6. Any disease or condition in which the use of the standard anti-TB drugs (or any of their components) are contraindicated. This includes, but is not limited to, allergy to any TB drug or their components.
7. In females: a positive urine pregnancy test result
8. Confirmed autoimmune disorders (e.g. systemic lupus erythematosus)

Additional Exclusions for Gadolinium contrasted CMR

1. Any implanted devices that are not MR compatible (e.g. pacemaker, defibrillators, cerebral aneurysm clips, cochlear implants etc.)
2. Claustrophobia
3. Gadolinium allergy
4. Inability to lie on a flat surface for prolonged periods of time (e.g. severe congestive cardiac failure)
5. Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Drug exposure in PCF and mediates in Mtb load | 72 hours and 52 weeks
  To determine whether higher dose rifampicin (35mg/kg) increases pericardial fluid (AUC) RIF levels and increases time to positivity of mycobacterial culture at 72 hours compared to standard dose Rifampicin

SECONDARY OUTCOMES:
Mortality between study arms | week 8 and 52 weeks
  To investigate clinical outcome by mortality (attributable to PCTB and all cause)
re-accumulation of pericardial effusion between study arms | 52 weeks
  To investigate clinical outcome by comparing clinical evidence of constrictive pericarditis between study arms
TB-IRIS between study arms | 52 weeks
  To investigate clinical outcome by comparison of the incidence of TB immune reconstitution inflammatory syndrome (TB-IRIS) between study arms
Constrictive pericarditis between the study arms | 52 weeks
  Comparison of the incidence of constrictive pericarditis between the study arms
CMR evidence | 52 weeks
  To investigate clinical outcome by evidence on week 52 CMR of:
  1. Constrictive physiology
  2. Pericardial inflammation
  3. Pericardial thickening
  4. Pericardial fibrosis
  5. Inflammatory exudative or hemorrhagic pericardial effusion

OTHER OUTCOMES:
To investigate the safety and tolerability of RIF35 for PCTB by: | week 8 and 52 weeks
  1. The occurrence of Grade 3 or 4 transaminitis during ATT
  2. Permanent discontinuation of the RIF10 or RIF35 ATT arm at week 8
Discontinuation rate | 52 weeks
  Comparison of discontinuation rates between study arms Comparison of discontinuation rates between study arms
Change in Mtb bacterial load | 72 hours
  To investigate early change in Mtb bacterial load by measures other than culture TTP (CFU, Xpert ct values, ddPCR, CEQ, Mtb RNA, FujiLAM) in PCF over 72 hours by treatment allocation
Relationships between pericardial Mtb-specific T cells with Mtb bacterial load | 52 weeks
  To determine relationships between pericardial Mtb-specific T cells with Mtb bacterial load, treatment response and outcome in PCTB
Mtb-induced markers of host cell death pathways and Mtb bacterial load in PCTB | 52 weeks
  To assess whether there is association between Mtb-induced markers of host cell death pathways and Mtb bacterial load in PCTB

CONTACTS AND LOCATIONS:
Overall Officials: Mpiko U Ntsekhe, Professor, Principal Investigator — Department of Cardiology, Groote Schuur Hospital
Locations (2):
- South Africa (2):
  - Nelson Mandela Academic Hospital, Mthatha, Eastern Cape
  - Groote Schuur Hospital, Cape Town, Western Cape

IPD SHARING:
Plan to Share IPD: Undecided